CLINICAL TRIAL: NCT03399474
Title: Comparison of Analgesic Efficacy of Two Different Doses of Dexmedetomidine as Adjuncts to Lidocaine for Intravenous Regional Anesthesia: Randomized Clinical Trial.
Brief Title: Analgesic Efficacy of Two Doses of Dexmedetomidine as Adjuncts to Lidocaine for Intravenous Regional Anesthesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ghada Mohammed AboelFadl, Principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Assiut University Anathesia
Record Dates: First submitted 2017-12-21; First posted 2018-01-16 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Limb Deformity
Keywords: Regional Anesthesia, Dexmedetomidine and lidocaine
MeSH Terms: interventions — Lidocaine; Dexmedetomidine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lidocaine only (Active Comparator): Lidocaine intravenous in a dose of 3 mg/kg lidocaine 0.5% diluted in 40 ml isotonic saline for intravenous regional anesthesia.
  Interventions: Drug: Lidocaine Hydrochloride 2%
- 0.5 ug/kg dexmedetomidine (Experimental): Lidocaine intravenous in a dose of 3 mg/kg lidocaine 0.5% diluted in 40 ml isotonic saline (maximum dose200 mg)+ Dexmedetomidine intravenous in a dose of 0.5 ug/kg, with the total volume diluted to 40 ml with normal saline 0.9%. The solution will be injected at a rate of 20 ml/min for intravenous regional anesthesia.
  Interventions: Drug: Dexmedetomidine 0.5 ug/kg
- 0.25 ug/kg dexmedetomidine (Experimental): 1 Lidocaine intravenous in a dose of 3 mg/kg lidocaine 0.5% diluted in 40 ml isotonic saline (maximum dose200 mg)+ Dexmedetomidine intravenous in a dose of 0.25 ug/kg, with the total volume diluted to 40 ml with normal saline 0.9%. The solution will be injected at a rate of 20 ml/min. for intravenous regional anesthesia.
  Interventions: Drug: Dexmedetomidine Injection 0.25 ug/kg

INTERVENTIONS:
Drug: Lidocaine Hydrochloride 2% — Lidocaine Hydrochloride 2%
  Arms: Lidocaine only
Drug: Dexmedetomidine 0.5 ug/kg — pecedex
  Arms: 0.5 ug/kg dexmedetomidine
Drug: Dexmedetomidine Injection 0.25 ug/kg — pecedex
  Arms: 0.25 ug/kg dexmedetomidine

SUMMARY:
Intravenous Regional Anesthesia (IVRA) was first used by August Bier in 1908. This technique is easy to administer, reliable and cost-effective for short surgical procedures of the extremities performed on an ambulatory basis with success rate of approximately 95% - 100% .

Lidocaine becomes the local anesthetic of choice for Intravenous Regional Anesthesia (IVRA) because of the lack of cardiac toxicity and neurotoxicity. But, delayed onset of action, poor muscle relaxation and lack of postoperative analgesia are the major limitations of this technique. Accordingly, many additives have been tried to overcome this problem. Muscle relaxants, ketamine,ketorolac, clonidine and opioids are examples of these adjuvants, and their effects have been studied in detail.

An ideal anesthetic agent for IVRA should have rapid analgesic effect to reduce tourniquet pain and its effects should last longer enough after deflating tourniquet. To achieve this, other drugs including narcotics, nonsteroidal anti-inflammatory drugs, ketorolac, clonidine, nitroglycerin (TNG), dexmedetomidine, magnesium, and neostigmine were used in combination with lidocaine in different studies. This study aims 1- To compare the anesthetic and analgesic efficacy of Dexmedetomidine and lidocaine versus lidocaine only during IVRA (Bier's block) and 2-To compare anesthetic and analgesic efficacy of different doses of dexmedetomidine when used as adjuvants to lidocaine during IVRA (Bier's block).

DETAILED DESCRIPTION:
Preoperative evaluation of the patients will be done including medical history, physical examination, and laboratory investigations. Patients should be in fasting state for at least 8 h before surgery, and the visual analog scale (VAS) (from 0 to 10: 0 = no pain up to 10 = severe pain) will be explained to the patients to express their pain.

On arriving at the operating room, routine intraoperative monitors will be applied, such as a noninvasive blood pressure monitor, a five-lead ECG, and a pulse oximeter. Two (20 G) venous cannulae will be inserted, one in the dorsum of the operative hand and one in the other hand, for fluid infusion during surgery and for any intravenous medications.

Patients will be premedicated with IV 0.05 mg/Kg of midazolam. After the patient is taken to the operating room, mean arterial blood pressure (MAP), peripheral oxygen saturation (SPO2) and heart rate (HR) will be monitored. The operative arm will be elevated for 2 minutes then exsanguinated with an esmarch bandage. A pneumatic double tourniquet will be placed a round upper arm, and the proximal cuff will be inflated to 250 mmHg. Circulatory isolation of the arm will be verified by inspection, absence of radial pulse, and loss of pulse oximetry tracing in the ipsilateral index finger. After the bandage is removed, 40 ml of the respective solutions will be injected over 20 seconds by an anesthesiologist.

The Sensory block will be assessed by pinprick performed with a 22-gauge needle every 30 seconds until the dermatomal sensory block of medial and antebrachial cutaneous, ulnar, median and radial nerves achieved. Motor function will be assessed by asking the patients to flex and extend his/her wrist and fingers and complete motor block will be noted when no voluntary movement is possible. Sensory block onset time will be noted as the time elapsed from drug injection to complete sensory block achieved in all dermatomes. Motor block onset time is the time elapsed from injection of study drug to complete motor block. After complete sensory and motor blocks is achieved, the distal tourniquet will be inflated to 250 mmHg, and the proximal tourniquet will be released and the surgery will be s started.

MAP, HR and SPO2 level will be recorded before application of tourniquet and after the application of tourniquet every five minute and were measured after release of the tourniquet, and postoperatively at 30 min, 1 hr, 2 hr, 3 hr, 4 hr, 6 hr and 24 hours. Pain due to the tourniquet will be ssessed with visual analogue scale (VAS) scores (0 = no pain and 10 = worst pain imaginable).

Levels of sedation will be assessed with the Ramsey sedation scale as follows: 1-patient is anxious and agitated or restless or both, 2-patients is cooperative, oriented and tranquil, 3-patient responds to command only, 4-patient exhibits brisk response to light glabellar tap or loud auditory stimulus, 5-patient exhibits a sluggish response to light glabellar tap or loud auditory stimulus, and 6-patients exhibits no response .

Both VAS and sedation levels will be recorded before and after the application of tourniquet and during the operation (10, 15, 20, 30, 40, 50 and 60 min). When pain due to tourniquet was > 3 on the VAS, patients will be given nalbuphine 5 mg intravenously increments up to 0.1 mg/kg and total administered dose will be noted.

Oxygen will be administered with face mask if SPO2 is lower than 91%.

At the end of the operation patients will be asked to qualify the operative conditions such as tourniquet pain or incisional pain.

The tourniquet will be not deflated before 30 min and was not inflated more than 1.5 hours. At the end of the operation, the tourniquet deflation will be performed by cyclic deflation technique (the tourniquet was deflated three times in a cyclic manner with 10 seconds period of deflation).

Sensory recovery time will be documented (time elapsed after tourniquet deflation up to recovery of pain in all innervated areas determined by pinprick test).

Motor block recovery time will be noted (the time elapsed after tourniquet deflation up to movement of fingers). Also, first analgesic requirement time will be noted (the time elapsed after tourniquet release to the first patient request of analgesic).

In the postoperative period if patients starts to complain (VAS > 3); rescue analgesia will be given in the form of paracetamol (Perfalgan®) 1gm IV drip and/or diclofenac sodium (Voltaren®) 75 mg IM, and/or nalbuphine 5 mg IV (with maximum daily dose of 2 mg/Kg/day) till VAS ≤ 3.And total amount of nalbuphine administered in first 24 hours to each group will be recorded.

During the first 2 hours in the post-anesthetic care unit and later in the surgical ward, patients will be questioned for circumoral numbness and tingling, nausea and vomiting, skin rash, tinnitus, gastric discomfort and other side effects are noted if encountered and MAP, HR and VAS scores will be assed every 2 hours postoperatively during the first 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 20-60 years with American society of anesthesiologists physical status I or II undergoing minor hand or forearm surgeries (duration of surgery 60 min or less, such as carpal tunnel release, ganglion excision, trigger finger, tendon or nerve repair, and fracture finger or metacarpal bone) .

Exclusion Criteria:

* Patients with Raynaud's disease,
* history of drug allergy, sickle cell anemia, Liver diseases and kidney diseases
* Patients who had a history of allergy to the drugs used, recent or chronic use of analgesics,
* uncontrolled hypertension, diabetic neuropathy, peripheral ischemia, , or any psychological disturbances

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
The time to first analgesic request. | 24 hours
  if patients starts to complain (VAS > 3); rescue analgesia will be given in the form of paracetamol (Perfalgan®) 1gm IV drip and/or diclofenac sodium (Voltaren®) 75 mg IM, and/or nalbuphine 5 mg IV (with maximum daily dose of 2 mg/Kg/day) till VAS ≤ 3.And total amount of nalbuphine administered in first 24 hours to each group will be recorded.

SECONDARY OUTCOMES:
Pain due to the tourniquet assessed with visual analogue scale (VAS) scores before and after the application of tourniquet and during the operation | 24 hours
  Pain due to the tourniquet will be ssessed with visual analogue scale (VAS) scores (0 = no pain and 10 = worst pain imaginable).
Levels of sedation assessed with the Ramsey sedation scale before and after the application of tourniquet and during the operation | 24 hours
  Levels of sedation will be assessed with the Ramsey sedation scale as follows: 1-patient is anxious and agitated or restless or both, 2-patients is cooperative, oriented and tranquil, 3-patient responds to command only, 4-patient exhibits brisk response to light glabellar tap or loud auditory stimulus, 5-patient exhibits a sluggish response to light glabellar tap or loud auditory stimulus, and 6-patients exhibits no response .
The onset, duration times of both sensory and motor blocks, Sensory block onset time, Motor block onset time | 24 hours
  Sensory block onset time will be noted as the time elapsed from drug injection to complete sensory block achieved in all dermatomes. Motor block onset time is the time elapsed from injection of study drug to complete motor block.

CONTACTS AND LOCATIONS:
Locations (1):
- Ghada M Ab Elfadl, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided